CLINICAL TRIAL: NCT01493544
Title: Prevalence Study and Regular Practice (Diagnosis and Treatment) Among General Practitioners in Populations at Risk of COPD in Latin America
Brief Title: Prevalence Study and Regular Practice Among General Practitioners in Populations at Risk of Chronic Obstructive Pulmonary Disease (COPD) in Latin America
Acronym: PUMA PROJECT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RLA-XXX-2011/1
Record Dates: First submitted 2011-12-12; First posted 2011-12-16 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; smokers; primary care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
PUMA is an observational, multicentre, multinational, cross-sectional study with primary care physicians (primary care, general and family physicians). Participants will be selected sequentially among patients at risk for Chronic Obstructive Pulmonary Disease (COPD) who attend primary care consultation (primary care, general and family physicians). The inclusion visit will be a regularly scheduled or spontaneous consultation for patients, and this appointment with the physician will not depend on the study. During the appointment, data will be collected from the patient and the physician.

DETAILED DESCRIPTION:
PREVALENCE STUDY AND REGULAR PRACTICE (DIAGNOSIS AND TREATMENT) AMONG GENERAL PRACTICIONERS IN POPULATIONS AT RISK OF COPD IN LATIN AMERICA

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged more or equal than 40
* Current or former smokers and/or patients exposed to biomass combustion:

Cigarettes: more or equal than 10 packs/year; Pipes: more or equal than 50 pipes/year; Cigars: more or equal than 50 cigars/year; Combustion: more or equal 100 hours/firewood/year

Exclusion Criteria:

* Pregnancy
* Patients with contraindications for spirometry
* Physical or mental disability rendering the patient unable to undergo a spirometry test and to contribute data to the study
* Heart rate ≥ 120 beats by minute
* Patients currently undergoing treatment for tuberculosis
* A patient who is participating in an interventional clinical trial or was previously included in this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 40 or more, smokers or former smokers and/or people exposed to biomass combustion, who attend primary care consultation.
Sampling Method: Non-Probability Sample
Enrollment: 1907 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with an affirmative response to specific categories on the PUMA questionnaire. | Baseline
  PUMA Questionnaire: Based on the PLATINO questionnaire. Applied to patients to describe different aspects potentially related to Chronic Obstructive Pulmonary Disease (COPD) such as: respiratory symptoms, smoking, respiratory medication, health care resources usage, comorbidieties, etc., as well as the registration of procedures (spirometry and oximetry) carried out and anthropometric data.
FEV1 spirometry measures. | Baseline and visit 2 up to 4 weeks after baseline (if applicable)
  FEV1 is the volume of air expelled from the lungs in 1 second.
  The second visit will be scheduled only for those patients who do not meet criteria for deferring spirometry.
SaO2 (Arterial Oxygen Saturation) - pulse oximetry. | Baseline and visit 2 up to 4 weeks after baseline (if applicable)
  The second visit will be scheduled only for those patients who do not meet criteria for deferring spirometry.
Number of participants with an affirmative response to specific categories on the Medical History Questionnaire (if applicable). | Baseline
  Questionnaire based on the patient's personal medical history at the site. Its application will be subject to the existence of a prior medical history for the patient at site. If the patient has no prior medical history at site, then this questionnaire will not apply.
FEV1/FVC spirometry measures. | Baseline and visit 2 up to 4 weeks after baseline (if applicable)
  Ratio of Forced Expiratory Volume in 1 second (volume of air expelled from the lungs in 1 second) by the Forced Vital Capacity (FVC, the volume of air that can forcibly be blown out after full inspiration) is a spirometric measure (lung function test) used to demonstrate airway obstruction.
  The second visit will be scheduled only for those patients who do not meet criteria for deferring spirometry.
Heart rate (HR) - pulse oximetry. | Baseline and visit 2 up to 4 weeks after baseline (if applicable)
  The second visit will be scheduled only for those patients who do not meet criteria for deferring spirometry.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Montes de Oca, Internist - Pulmonologist, Study Chair — Universidad Central de Venezuela
Locations (18):
- Argentina (7):
  - Research Site, Belén de Escobar, Buenos Aires
  - Research Site, Ezeiza, Buenos Aires
  - Research Site, Los Polvorines, Buenos Aires
  - Research Site, Martínez, Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Ramos Mejía, Buenos Aires
  - Research Site, Capital Federal, Buenos Aires F.D.
- Colombia (5):
  - Research Site, Medellín, Antioquia
  - Research Site, Barranquilla, Atlántico
  - Research Site, Manizales, Caldas Department
  - Research Site, Armenia, Quindío Department
  - Research Site, Cali, Valle del Cauca Department
- Research Site, Montevideo, Montevideo Department, Uruguay
- Venezuela (5):
  - Research Site, Barquisimeto
  - Research Site, Caracas
  - Research Site, Maracaibo
  - Research Site, Porlamar
  - Research Site, Valencia

REFERENCES:
- [Derived] Lopez Varela MV, Montes de Oca M, Rey A, Casas A, Stirbulov R, Di Boscio V; PUMA Team. Development of a simple screening tool for opportunistic COPD case finding in primary care in Latin America: The PUMA study. Respirology. 2016 Oct;21(7):1227-34. doi: 10.1111/resp.12834. Epub 2016 Jun 20. PMID 27319305